CLINICAL TRIAL: NCT06811584
Title: Peanut Ball in Labor to Reduce Anxiety and Pain: Single-blind Randomized Clinical Trial
Brief Title: Peanut Ball in Labor to Reduce Anxiety and Pain
Acronym: BAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ricardo A Gutierrez Ramirez, MD, MSc, FACOG (Other)
Responsible Party: Sponsor-Investigator, Ricardo A Gutierrez Ramirez, MD, MSc, FACOG, Titular professor, Universidad Nacional Autonoma de Honduras
Organization: Universidad Nacional Autonoma de Honduras (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: PGO-UNAH-48-7-2025
Record Dates: First submitted 2025-01-31; First posted 2025-02-06 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Labor Stage, First; Anxiety; Pain Intensity Assessment
Keywords: Peanut ball; Labor stage, first; anxiety; pain intensity assesment
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Single-blind, parallel-group, efficacy, superiority, single-blind clinical trial.
Who Masked: Outcomes Assessor
Masking Description: Both the patient and the principal investigator will know the intervention, the data analyst researcher does not know the group to which the patients have been assigned.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Peanut ball (Experimental): Participants will be provided with a peanut ball, and she will be allowed to use it at least every two hours for a period of 30 minutes.
  Interventions: Device: Peanut ball
- Standard management (No Intervention): women will not use the peanut balloon and will receive standard care for labor, which may include measures such as pharmacologic pain relief and other labor management interventions.

INTERVENTIONS:
Device: Peanut ball — Participants will be provided with a mani ball, which will be covered by a cover provided by the investigator. This cover will be changed for each patient. The ball will be placed between the participant's knees, and she will be allowed to use it at least every two hours for a period of 30 minutes. Participants will also have the option to use the balloon more frequently if they wish. Balloon use will be discontinued when the cervical os reaches 10 cm dilation or when the participant is ready to begin the pushing process.
  * The positions to be performed with the peanut ball will be:
  * Side lying
  * Bent position
  * Semi-sitting position
  * Taylor position.
  Other Names: peanut shaped ball; peanut labor ball
  Arms: Peanut ball

SUMMARY:
An open clinical trial-type study of randomized assignment groups, an interventional model of parallel assignment, will be carried out to establish whether or not there are significant differences in the levels of anxiety and intensity of pain, in labor in patients who use the peanut ball and those that don't.

DETAILED DESCRIPTION:
The process of labor is a unique and significant experience in a woman's life, and obstetric care is constantly seeking strategies to effectively improve the experience of this crucial event.

Now in response to the growing global attention to quality and respect in maternity care, the International Childbirth Initiative (ICI) has outlined "12 steps to safe and respectful maternity care, which advocate for safe and respectful maternity care".

The declaration of rights of the World Health Organization (WHO) in the year 2021 highlights the urgency of "acting now for a safe and respectful childbirth", reinforcing the global commitment to respect, protect and fulfill the right to health, particularly maternal health. In this context, it emphasizes the need to ensure a positive, satisfactory and well-being experience during pregnancy and childbirth, in Honduras is part of this group of initiatives in order to promote an environment of respect for the mother at the time of childbirth.

Most healthy women can give birth with a minimum of medical procedures without putting at risk the mother-child binomial, the safest delivery is the one that evolves spontaneously and in which there is no unnecessary intervention, for that is necessary health facilities that have the requirements to provide delivery care and professionals who understand what are the basic needs of women during this physiological process. For decades, peanut balls have been used as a non-pharmacological complement for labor management. So far, this non-drug strategy has shown significant advantages in several aspects, among them, pain control, anxiety reduction, improvement in maternal experience and positive influence on obstetric indicators.

In the national and international context of guidelines and commitments towards safe and respectful maternal care, there is a need for a localized and specific evaluation of interventions, such as the use of the peanut balloon, to understand its efficacy in reducing anxiety and pain during labor, With the development of this study we aim to evaluate the efficacy of the use of the peanut balloon as a therapeutic intervention to reduce anxiety and pain in women during labor at Hospital Escuela Universitario in the period from June 2024 to June 2025, which could contribute to the knowledge about therapeutic practices in the obstetric context, providing solid scientific evidence on the efficacy of the use of the peanut balloon. The successful implementation of this intervention could have a positive impact on both women's experience and obstetric clinical practice, and is expected to serve to establish a protocol for the management of labor and delivery using the peanut ball.

ELIGIBILITY:
Inclusion Criteria:

* Submission of a signed and dated informed consent form.
* Declared willingness to comply with all study procedures and availability for the duration of the study.
* Female 18 to 45 years of age
* USG having normal amniotic fluid index and monitoring.
* Gestational age > 36 weeks 0 days
* Singleton pregnancy
* Cephalic presentation.
* Nulliparous
* Cervical dilatation less than 5 cm
* Spontaneous evolution
* Induction or conduction of labor

Exclusion Criteria:

* Pre-pregnancy BMI >30 kg/m2 or obesity
* Multiple gestation
* Intrauterine fetal death
* Musculoskeletal problems that hinder ball use
* Receiving magnesium sulfate
* Premature rupture of the membrane greater than 24 hours
* Cervical incompetence
* High risk pregnancies (Preeclampsia/eclampsia, cholestasis, intrauterine growth retardation, fetal anomaly, polyhydramnios or oligohydramnios, heart disease, HIV).
* Labor dystocia
* Diagnosis of mental illness.
* Multiparous.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 163 (Actual)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-09-01 (Actual)

PRIMARY OUTCOMES:
anxiety level | Since intervention until 8 hours
  Pain Anxiety Symptom Scale - Short Format 20 (PASS-20), This test measures 20 items using a Likert scale from 1 to 5, with a minimum score of 20 and a maximum of 100.
Visual Analog Pain Scale | Since intervention until 24 hours
  It is a horizontal line of 10 centimeters, at the ends of which the extreme expressions of a symptom are shown. On the left side is located the absence or lower intensity and on the right side the higher intensity. The patient is then asked to mark on the line the point indicating the intensity and it is measured with a millimeter ruler. The intensity is expressed in centimeters or millimeters

SECONDARY OUTCOMES:
Maternal Well-being in Childbirth Scale 2 (BMSP2) | Since intervention until 24 hours
  The total scale score defines three levels of maternal well-being: excellent (score > 200), adequate (score > 183 and <. 200), and poor (score < 183), the score range has a minimum of 47 and a maximum of 235
The Wijma Delivery Expectancy/Experience Questionnaire (W-DEQ) | Since intervention until 24 hours
  measures the Fear of childbirth. It is divided into 2 parts, part A with 32 items with a Likert scale (32 to 192 points) and part B with 30 points with a Likert scale (30 to 180 points)

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo A. Gutierrez Ramirez, MD, MSc., Study Director — Universidad Nacional Autonoma de Honduras
Locations (1):
- Hospital Escuela, Tegucigalpa, Francisco Morazán Department, Honduras

IPD SHARING:
Plan to Share IPD: No
It is not necessary, none of the 18 HIPAA identifiers will be placed

REFERENCES:
- [Background] Delgado A, Katz L, Melo RS, Amorim M, Lemos A. Effectiveness of the peanut ball use for women with epidural analgesia in labour: a systematic review and meta-analysis. J Obstet Gynaecol. 2022 Jul;42(5):726-733. doi: 10.1080/01443615.2021.1997959. Epub 2022 Jan 7. PMID 34996318